CLINICAL TRIAL: NCT01703871
Title: Music During Diagnostic Hysteroscopy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Cafa Ester Valentina, medical doctor, Campus Bio-Medico University
Other Study IDs: HM-1
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-09

CONDITIONS: Pain; Anxiety; Tolerability
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Office Hysteroscopy is associated with a level of anxiety that could condition tolerability of the procedure by the patient.

The aim of this study is to evaluate the impact of music on anxiety state, expected and received pain by patients during office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for office hysteroscopy in menopausal status or in childbearing age

Exclusion Criteria:

* Previous diagnostic hysteroscopy and/or RCU
* Current or recent pelvic Inflammation
* Invasive cervix cancer
* Ongoing pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-09